CLINICAL TRIAL: NCT01491139
Title: A Phase I/II Study of Olaparib in Addition to Cisplatin Based Concurrent Chemoradiotherapy for Patients With High Risk Locally Advanced Squamous Cell Carcinoma of the Head and Neck (HNSCC)
Brief Title: Phase I Study of Olaparib With Cisplatin Based Chemoradiotherapy in Squamous Cell Carcinoma of the Head and Neck
Acronym: ORCA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped due to issues surrounding development and formulation of olaparib
Sponsor: University College, London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-023599-24; 62346992 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Radiotherapy; Biomarkers, pharmacological; Pharmacokinetics; Genetic Markers; Cisplatin; Poly(ADP-ribose) Polymerases; AZD 2281; Radiotherapy, Intensity-Modulated; Head and Neck; Chemoradiotherapy; SCC
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — olaparib; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): All patients will receive induction chemotherapy (cisplatin and 5-FU), followed by cisplatin chemotherapy and radiotherapy in addition to oral olaparib.
  Induction chemotherapy (21 day cycle)
  * Drug: cisplatin 80mg/m2 (day 1)
  * Drug: 5-FU (fluorouracil) 1000mg/m2/day (day 1-4 continuous infusion)
  olaparib plus chemoradiotherapy (8 weeks)
  * Drug: olaparib
  * Drug: Cisplatin
  * Radiation
  Interventions: Drug: olaparib; Drug: cisplatin; Radiation: Intensity Modulated Radiotherapy

INTERVENTIONS:
Drug: olaparib — Given twice daily. Exposure will escalate by daily dose and duration.
  Other Names: AZ2281
Drug: cisplatin — Dose will be 35mg/m2 i.v. once weekly.
Radiation: Intensity Modulated Radiotherapy — Total dose will be 70Gy in 35 fractions over 7 weeks.

SUMMARY:
The aim of this study is to find the safe dose and best dosing schedule of olaparib to give in combination with cisplatin based chemoradiotherapy (CRT) in patients with locally advanced head and neck cancer. The dose decided on in this part of the study will become the recommended dose for the randomised Phase II trial.

DETAILED DESCRIPTION:
This is a dose escalating Phase I/II trial evaluating the safety and tolerability of the addition of olaparib to CRT in high risk locally advanced human papillomavirus (HPV) negative Squamous Cell Carcinoma of the Head and Neck (HNSCC). A fixed dose of weekly cisplatin and intensity-modulated radiation therapy (IMRT) will be used, with doses of olaparib escalating for consecutive days and both dose level and duration will be increased through each cohort.

This Phase I trial will assess how olaparib, a poly ADP ribose polymerase (PARP) inhibitor is tolerated when added to standard chemoradiotherapy treatment.

Patients will be recruited from sites in the UK only.

A placebo controlled, randomised Phase II trial will follow once the recommended dose and schedule of olaparib has been established.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high risk, locally advanced HNSCC patients (TNM staging: T-any N2/3 M0, bulky T3 or T4 N-any M0) who would normally be offered cisplatin-based radical chemoradiotherapy
* Estimated life expectancy of at least 12 weeks
* WHO performance status of 0 or 1
* Aged ≥18 years of age
* Adequate major organ function
* Willing to use contraception for the duration of the trial treatment and for six months after completion of treatment
* Able to give informed consent
* Willing and able to comply with the protocol for the duration of the study

Exclusion Criteria:

* Head & neck cancers of the following types:
* Nasopharyngeal and paranasal sinus tumours,
* Oral squamous cell carcinomas (tumours of the oral cavity),
* Human Papilloma Virus positive oropharyngeal tumours (tonsillar and tongue base tumours)
* Confirmed distant metastatic disease
* Previous chemotherapy or radiotherapy for the treatment of HNSCC tumour
* Previous therapy with a PARP inhibitor
* Pre-existing gastrointestinal disorders that may interfere with the delivery or absorption of olaparib
* Grade 3 or 4 peripheral neuropathy
* Significant hearing difficulties or tinnitus (deaf patients can be included)
* The current use of drugs which are known to inhibit or induce CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Frequency of dose limiting toxicities | 6 weeks post completion of treatment

SECONDARY OUTCOMES:
Complete response rate | 12 weeks post completion of treatment
Time to loco-regional progression | 2 years post completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Martin D Forster, MBBS, Principal Investigator — University College London Hospitals